CLINICAL TRIAL: NCT01545219
Title: A Double-blind, Placebo-controlled, Randomized Crossover Study to Determine the Effects of Xylooligosaccharides (XOS), B. Lactis (BI07) and XOS + BI07 Upon the Gut Microbiota and Immune Response of Healthy Volunteers
Brief Title: A Study of a Prebiotic, a Probiotic and a Synbiotic Upon the Gut Microbiota and Immune Response of Healthy Volunteers
Acronym: XOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Danisco (Industry)
Responsible Party: Principal Investigator, Caroline Childs, Post doctoral research fellow, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 08/38
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Gut Microbiota; Bowel Function; Immune Function; Plasma Lipids
MeSH Terms: interventions — Prebiotics; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prebiotic (Experimental)
  Interventions: Dietary Supplement: Prebiotic
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Bi-07
- Synbiotic (Experimental)
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — 8g/day xylo-oligosaccharide
  Arms: Prebiotic
Dietary Supplement: Bi-07 — 10^9 CFU B. lactis / day
  Arms: Probiotic
Dietary Supplement: Synbiotic — 8g/day xylo-oligosaccharide + 10^9 CFU Bi-07
  Arms: Synbiotic
Dietary Supplement: Placebo — 8g/day maltodextrin
  Arms: Placebo

SUMMARY:
Healthy volunteers will be recruited to a study where they will be given four different treatments over a 28 week period. These treatments include: a prebiotic, a probiotic, a synbiotic (prebiotic + probiotic) and a placebo. Faecal samples, blood and saliva will be collected and analysed for changes in faecal microbial populations and selected immune responses.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of XOS (administered at 8g/day), B. lactis BI07 (administered at 109 CFU/day) and the synbiotic combination of both (8g/day XOS and 109 CFU/day B. lactis BI07) on the human gut microbiota.

A double-blind, placebo-controlled, randomized crossover study will be conducted in 44 healthy volunteers. The placebo will be maltodextrin (a food grade ingredient, administered at 8g/day).

Changes in the gut microbiota will be determined by measuring bacterial population levels in human faeces using fluorescence in situ hybridisation (FISH) with 16S rRNA targeted oligonucleotide probes. Concentrations of short chain fatty acids (SCFA) will be quantified using gas chromatography (GC).

In addition to analyses performed on the samples at the University of Reading, analyses on microbial metabolites and selected members of the microbiota will also be performed at Danisco Finland, Kantvik. University of Reading will therefore provide Danisco Kantvik with faecal samples of appropriate size.

The secondary objective of this study is to examine the effects of XOS (8g/day), B. lactis BI07 (109 CFU/day) and the synbiotic (8g/day of XOS and 109 CFU/day of B. lactis BI07) on bowel function, immune function and plasma lipids in 44 healthy volunteers. This will be achieved using volunteer diaries of bowel function and mood, and by investigating total plasma lipids, mucosal immunity (salivary and faecal IgA), total leukocyte numbers, expression of cell surface markers on immune cells to identify cell subsets and activation markers, production of inflammatory markers by whole blood cultures, plasma chemokines, phagocytosis and oxidative burst by monocytes and granulocytes, plasma/serum immunoglobulins, acute phase proteins, complement proteins and soluble adhesion molecules.

ELIGIBILITY:
Inclusion Criteria:

* signed consent form
* age 25-65 years
* body mass index 20-30 inclusive
* good general health as determined by medical questionnaires
* additional inclusion criteria: as far as possible, target volunteer group will have mild constipation (bowel movement of less than 1/day, hard stool consistency)

Exclusion Criteria:

* • Evidence of physical or mental disease or planned major surgery, which might limit participation in or completion of the study

  * History of drug abuse, including alcohol
  * Severe allergy or a history of severe abnormal drug reaction
  * Participation in experimental drug trial within four weeks prior to study
  * Participation in prebiotics or laxative trial within the previous three months
  * Use of antibiotics within the previous six months
  * Chronic constipation, diarrhoea or other chronic gastro-intestinal complaint
  * Intake of other prebiotics or probiotics, drugs active on gastrointestinal motility, or a laxative of any class for four weeks prior to study
  * Use of prescribed medication
  * Regular use of aspirin or other anti-inflammatory drugs

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Changes to the gut microbiota | 7 months
  Changes in faecal bacterial populations will be assessed through the use of FISH with molecular probes targeting 16S rRNA genes. Genotypic probes targeting the predominant components of the gut microflora (Bacteroides, Bifidobacterium, Clostridium, Lactobacillus, Eubacterium, Atopobacterium, Streptococcus, sulphate reducing bacteria and enterobacteria) and total bacteria will be tagged with fluorescent markers such that quantifiable changes may be determined. Concentrations of short chain fatty acids (SCFA) will be quantified using gas chromatography (GC).

SECONDARY OUTCOMES:
Bowel function, immune function and plasma lipids | 7 months
  This will be achieved using volunteer diaries of bowel function and mood, and by investigating total plasma lipids, mucosal immunity (salivary and faecal IgA), total leukocyte numbers, expression of cell surface markers on immune cells to identify cell subsets and activation markers, production of inflammatory markers by whole blood cultures, plasma chemokines, phagocytosis and oxidative burst by monocytes and granulocytes, plasma/serum immunoglobulins, acute phase proteins, complement proteins and soluble adhesion molecules.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn R Gibson, BSc, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom